CLINICAL TRIAL: NCT03175588
Title: Comparison of Effects of Interactive Video Games and Activity Based Approaches on Mobility and General Well Being in the Elderly
Brief Title: Comparison of Effects of Interactive Video Games in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Aynur CICEK, PT, MSc, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08.02.2017 / 52639
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Virtual Rehabilitation
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: There will be three groups in this study. Two intervention and one control gruop to be compared after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual rehabilitation (Experimental): video based exercise
  Interventions: Other: Virtual Rehabilitation
- physical Activity (No Intervention): different type of physical Activity

INTERVENTIONS:
Other: Virtual Rehabilitation — Nintendo Wii program with balance board, which is the most frequently preferred game consoles in rehabilitation will be used
  Arms: virtual rehabilitation

SUMMARY:
The aim of this study is to assess the effectiveness of interactive video-games on mobility and wellbeing and to compare them with activity-based approaches in geriatric population.

100 people living in Bahcelievler nursing home will be evaluated and volunteers who meet the criteria will be included in the study. Persons will be placed in the study groups in consideration of their interests. One group will be included in Nintendo Wii program with balance board, which is the most frequently preferred game consoles in rehabilitation, and video-games will run for 30 minutes two days a week for 8 weeks. The other group will participate a program consisting of various physical activities for the same duration; The results of both groups will be compared with a control group.

DETAILED DESCRIPTION:
100 people living in Bahcelievler nursing home will be evaluated and volunteers who meet the criteria will be included in the study. Persons will be placed in the study groups in consideration of their interests. One group will be included in Nintendo Wii program with balance board, which is the most frequently preferred game consoles in rehabilitation, and video-games will run for 30 minutes two days a week for 8 weeks. The other group will participate a program consisting of various physical activities for the same duration; The results of both groups will be compared with a control group.

ELIGIBILITY:
Inclusion Criteria:

* mini mental test score abowe 21 age between 65 and 85

Exclusion Criteria:

neurological disorders orthopedical problems

-

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 58 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-03-11 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 5 minute
  Balance measurement

SECONDARY OUTCOMES:
10-meter walking test | 3 minute
  functional ability and balancing
WHQOL-Bref | 15 minute
  quality of life
Hamilton Depression Scale | 15 minute
  Assessment of emotional situation

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Razak Ozdincler, Prof, Study Director — Istanbul University
Locations (1):
- Bahcelievler Community dwelling, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No